CLINICAL TRIAL: NCT00190827
Title: The Effectiveness of Duloxetine Compared With Placebo in the Treatment of Predominant Stress Urinary Incontinence
Brief Title: Effectiveness of Duloxetine in the Treatment of Stress Urinary Incontinence(Uncontrolled Leakage of Urine)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6195; F1J-MC-SBBR
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine
Drug: placebo

SUMMARY:
The study evaluates the effectiveness of duloxetine in reducing urinary incontinence occurrences in women due to physical stress(e.g. stomach pressure on bladder). Incontinence is the inability to control bladder function with leakage of urine.

ELIGIBILITY:
Inclusion Criteria:

* female outpatients > or = 18 years of age
* experience episodes of stress urinary incontinence
* must have an educational level and degree of understanding English
* are free of urinary tract infections
* can use the toilet independently

Exclusion Criteria:

* any in or outpatient surgery in the last six months
* suffer from severe constipation
* extension of any internal organs beyond vaginal opening
* currently breastfeeding
* any nervous diseases affecting normal urinary function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2003-09; Study Completion 2006-05

PRIMARY OUTCOMES:
Compare duloxetine 40 mg BID with placebo in the reduction of incontinence episode frequency(IEF). Study visits occur every two weeks in therapy phase.
Evaluate the effects of different regimens of dose escalation and tapering effects on incidence of most prevalent adverse events.

SECONDARY OUTCOMES:
Assessment of overall patient safety.
Reduction of IEFs using standardized instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559 or 1-317-615-4559) Monday-Friday 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559 OR 1-317-615-4559) Mon-Fri from 9am to 5pm Eastern time(UTC/GMT - 5 hours, EST) or speak with your personal physician, Rio de Janeiro, Brazil
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559 or 1-317-615-4559) Mon-Fri from 9am to 5pm Eastern time(UTC/GMT - 5 hours, EST) or speak with your personal physician, Québec, Quebec, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559 OR 1-317-615-4559) Mon-Fri from 9am to 5pm Eastern time(UTC/GMT - 5 hours, EST) or speak with your personal physician, Paris, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559 OR 1-317-615-4559) Mon-Fri from 9am to 5pm Eastern time(UTC/GMT - 5 hours, EST) or speak with your personal physician, Mainz, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559 OR 1-317-615-4559) Mon-Fri from 9am to 5pm Eastern time(UTC/GMT - 5 hours, EST) or speak with your personal physician, Torino, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559 OR 1-317-615-4559) Mon-Fri from 9am to 5pm Eastern time(UTC/GMT - 5 hours, EST) or speak with your personal physician, Mexico City, Mexico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559 OR 1-317-615-4559) Mon-Fri from 9am to 5pm Eastern time(UTC/GMT - 5 hours, EST) or speak with your personal physician, San Juan, Puerto Rico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559 OR 1-317-615-4559) Mon-Fri from 9am to 5pm Eastern time(UTC/GMT - 5 hours, EST) or speak with your personal physician, Barcelona, Spain